CLINICAL TRIAL: NCT06895044
Title: Evolution of Ocular Growth in Myopic Children: A Prospective Cohort Study
Acronym: PREMYOM1000
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SBN_2024_13
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ophtalmologic follow-up — alls exams included in ophtalmologic follow-up every 6 months for 5 years
Other: ophtalmological follow-up — all exams included in ophtalmological follow-up including axial length mesurment every 6 moths

SUMMARY:
Myopia and high myopia are the leading causes of visual impairment and blindness worldwide. The total number of myopic people globally was estimated to be 2.6 billion in 2020, and it could reach 4.8 billion by 2050 unless preventive interventions are implemented.

Strategies to slow the progression of myopia, such as contact lenses, orthokeratology, atropine, and increased time spent outdoors, have shown promising results, although evidence varies depending on the method. However, most research has been conducted in Asia, and there are few studies on ocular growth in myopic children in Europe. Meanwhile, the prevalence of myopia is also increasing significantly in Europe, particularly in France.

Understanding the growth of the myopic eye in European children is crucial. Cohort studies of myopic children are scarce and do not always include high-quality imaging. A cohort of myopic children with prospective collection of the best retinal and corneal images, along with ophthalmological exams to detail and model the growth of the myopic eye, will provide valuable insights to enhance our understanding of ocular growth and its inter-individual variability.

ELIGIBILITY:
Inclusion Criteria:

* Myopia in at least one eye, defined as a refractive error in spherical equivalent ≤ -0.50 diopters (autorefraction under cycloplegia)
* Affiliated or beneficiary of a social security system
* Explicit consent from a holder of parental authority

Exclusion Criteria:

* Presence of trauma in both eyes
* Presence of inflammatory conditions in both eyes
* History of intraocular surgery (cataract, filtering surgery, intra-vitreal surgery) in both eyes
* Patient benefiting from legal protection measures

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 6 to 17 years at inclusion, diagnosed with myopia (refractive error of -0.5 D or less in spherical equivalent in at least one eye)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2033-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
axial length | Year 5
  Measurement of axial length by IOL Master

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut Chapron, Dr, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France